CLINICAL TRIAL: NCT00456898
Title: A Randomized, Open-Label, 3-Period Crossover Study to Evaluate the Effect of Multiple Doses of DVS SR and Paroxetine on the CYP2D6 Biotransformation of Codeine to Morphine in Healthy Subjects.
Brief Title: Study Evaluating the Potential of DVS SR to Inhibit the CYP2D6 Pathway
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-1203
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Depressive Disorder, Major; Diabetic Neuropathies; Fibromyalgia; Vasomotor Symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Diabetic Neuropathies; Fibromyalgia | interventions — Paroxetine; Codeine

INTERVENTIONS:
Drug: desvenlafaxine sustained release (DVS SR)
Drug: Paroxetine
Drug: Codeine

SUMMARY:
To evaluate the effects of multiple oral doses of desvenlafaxine sustained release (DVS SR) and paroxetine on the biotransformation of codeine to morphine in healthy subjects. To assess the safety and tolerability of DVS SR and paroxetine when coadministered with codeine to healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, open-label, inpatient/outpatient, 3-period crossover study in healthy subjects.The study will consist of 3 treatment periods. In treatment period 1, subjects will be randomly assigned on study day 1. A single 60-mg dose of codeine will be administered to all subjects. In periods 2 and 3, subjects will receive either DVS SR 100 mg/day or paroxetine 20 mg/day until the steady state is reached. At steady state, subjects will receive codeine 60 mg concomitantly with either DVS SR 100 mg or paroxetine 20 mg, depending on the treatment sequence to which they are assigned. DVS SR 100 mg or paroxetine 20 mg administration will continue for an additional 2 days. In treatment period 3, subjects will receive the alternative treatment sequence.

ELIGIBILITY:
Inclusion criteria:

* Healthy men and nonlactating and nonpregnant women of nonchildbearing potential aged from 18 to 45 years.
* Body mass index in the range of 18 to 30 kg/m2 and body weight ≥50 kg.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history.

Exclusion criteria:

* History of bronchial asthma, of seizure disorder (other than a single childhood febrile seizure)and of any clinically important drug allergy and any known allergy to desvenlafaxine, venlafaxine, paroxetine, codeine, or any of the non-active excipients in the dosage forms.
* Use of any CYP2D6 inhibitors or inducers within 30 days before test article administration.
* Demonstration of a positive orthostatic test at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2007-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
the biotransformation of codeine to morphine and the safety and tolerability of DVS SR

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer